CLINICAL TRIAL: NCT07332026
Title: Evaluation of the Effect of Type 2 Diabetes Mellitus on the Success of Adult Pulpotomy
Acronym: controlled cli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Mohamed Sulaiman, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/6/2023
Record Dates: First submitted 2025-12-13; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Adult Pulpotomy Success in Diabetic Patients
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diabetic (Experimental): type 2 diabetic patients
  Interventions: Procedure: pulpotomy
- non-diabetic (Experimental): healthy patients
  Interventions: Procedure: pulpotomy

INTERVENTIONS:
Procedure: pulpotomy — complete excision of coronal pulp
Procedure: pulpotomy — excision of coronal pulp

SUMMARY:
The aim of the present study will be directed to evaluate the clinical and radiographic success of adult pulpotomies in type 2 diabetic and non-diabetic patients.

DETAILED DESCRIPTION:
Out of one hundred patients, Seventy Patients were selected from the outpatient clinic at the faculty of dental medicine Al-Azhar University to take part in this study. Diabetic and non diabetic patients aged between 30 and 65 years complaining of irreversible pulpitis related to the lower permanent first or second molar tooth . All patients were clinically reexamined and radiographically assessed using a periapical radiograph.

ELIGIBILITY:
lower first or second molar diagnosed with irreversible pulpitis in diabetic and non-diabetic patients

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Outcome assessment | 3, 6, 12 months
  Assessment of outcome was done using the technique described by Zanini et al. Each patient was evaluated at different time intervals;
  Treatment was considered successful if there was an intact final restoration, an asymptomatic tooth, and the periapical index score was 1.
  Treatment was considered Uncertain if the final restoration is intact, asymptomatic tooth, and the periapical index score of 2.
  Treatment was considered a failure if there was not an intact final restoration, irrelevant clinical symptoms and an irrelevant periapical index score.
  Treatment was considered a failure if there was an intact final restoration with symptoms and an irrelevant periapical index score.
  * Treatment was considered a failure if there was an intact final restoration, irrelevant clinical symptoms, and the periapical index was 3 or more.

CONTACTS AND LOCATIONS:
Locations (1):
- Moataz A AlKhawas, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided